CLINICAL TRIAL: NCT03386591
Title: Comparison of Naloxone Pharmacokinetics Using Marketed Naloxone Devices
Brief Title: Comparison of Naloxone Pharmacokinetics
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: Naloxone P1a-003
Record Dates: First submitted 2017-12-18; First posted 2017-12-29 (Actual); Last update posted 2018-03-09 (Actual); Status verified 2018-03

CONDITIONS: Opioid-use Disorder
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Naloxone; Syringes

STUDY DESIGN:
Intervention Model Description: This will be an inpatient open-label, randomized, 5-period, 5-treatment, 5-sequence, crossover study involving approximately 30 healthy subjects.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (5):
- Mucosal Atomization (1 administration) (Experimental): One Intranasal administration of 2 mL naloxone using a mucosal atomization device and syringe (1 mL/nostril)
  Interventions: Drug: Naloxone; Device: Mucosal atomization device and syringe
- Mucosal Atomization (2 administrations) (Experimental): Two Intranasal administrations of 2 mL naloxone using mucosal atomization device and syringe (1 mL/nostril) 2 minutes apart
  Interventions: Drug: Naloxone; Device: Mucosal atomization device and syringe
- Narcan 2mg (Experimental): One Intranasal administration of 2 mg naloxone using Narcan nasal spray
  Interventions: Drug: Naloxone; Device: Narcan
- Narcan 4mg (Experimental): One Intranasal administration of 4 mg naloxone using Narcan nasal spray
  Interventions: Drug: Naloxone; Device: Narcan
- Intramuscular auto injector (Experimental): One Intramuscular administration of 2 mg naloxone using Evzio auto-injector
  Interventions: Drug: Naloxone; Device: Intramuscular Auto Injector

INTERVENTIONS:
Drug: Naloxone — Comparing pharmacokinetics of naloxone
Device: Mucosal atomization device and syringe — Injection
  Arms: Mucosal Atomization (1 administration); Mucosal Atomization (2 administrations)
Device: Narcan — Nasal Spray
  Arms: Narcan 2mg; Narcan 4mg
Device: Intramuscular Auto Injector — Intramuscular injection
  Other Names: Evzio
  Arms: Intramuscular auto injector

SUMMARY:
Intranasal (IN) naloxone administration is an effective alternative to intravenous (IV) or intramuscular (IM) naloxone by emergency medical services for opioid overdoses and has been used successfully for this purpose as reported in clinical observational studies and a randomized controlled trial. Most of the published clinical studies concerning IN administration used an improvised kit of 2 mg naloxone/2 mL saline and a mucosal atomizer device (MAD), which is not FDA-approved for this indication. Pharmacokinetic (PK) data using these kits is not available in the published literature. This study is designed to determine the PK of naloxone following one and two IN administrations using the improvised kits compared to 2 and 4 mg delivered IN using the FDA-approved Narcan nasal spray device and 2 mg administered IM using the Evzio autoinjector.

ELIGIBILITY:
Inclusion Criteria:

* Males and females 18 to 55 years of age, inclusive
* Provide written informed consent
* BMI ranging from 18 to 32 kg/m2, inclusive
* Adequate venous access
* No clinically significant concurrent medical conditions determined by medical history, physical examination, clinical laboratory examination, vital signs, and 12-lead ECG
* Male subjects must agree to use an acceptable method of contraception with female partners as well as not to donate sperm from the screening visit until 90 days after the last study drug administration
* Female subjects of childbearing potential must agree to use an acceptable method of birth control from the start of screening until 30 days after the last study drug administration. Oral contraceptives are prohibited
* Agree not to ingest alcohol, drinks containing xanthine >500 mg/day (e.g., Coca Cola®, coffee, tea, etc.), or grapefruit/grapefruit juice or participate in strenuous exercise 72 hours prior to admission through the last blood draw of the study

Exclusion Criteria:

* Contact site directly for more information

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2018-01-03 (Actual); Primary Completion 2018-02-08 (Actual); Study Completion 2018-03-06 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic parameters of naloxone | 11 days
  Maximum plasma concentration, time of maximum observed concentration and area under the concentration-time curve

SECONDARY OUTCOMES:
Safety Assessments | 16 days
  Number of participants with AEs, vital signs, ECG, laboratory changes and nasal irritation following the administration of naloxone.

CONTACTS AND LOCATIONS:
Overall Officials: Debra Kelsh, MD, Principal Investigator — Vince and Associates Clinical Research
Locations (1):
- Vince and Associates Clinical Research, Overland Park, Kansas, United States

IPD SHARING:
Plan to Share IPD: No